CLINICAL TRIAL: NCT06075433
Title: A Prospective, Multicenter, Observational Study to Evaluate the Efficacy and Safety of 1 Year Duration of DAPT After GENOSS® DES Implantation in Patients with Coronary Artery Disease According to the Complex Higher-Risk Procedure
Brief Title: Efficacy and Safety of 1-year Duration of DAPT After GENOSS® DES Implantation in Patients with Coronary Artery Disease According to the Complex Higher-risk Procedure
Acronym: DAPTLong
Status: Recruiting | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS0501-14
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS Sirolimus Eluting Coronary Stent System: Patients with coronary artery disease treated with the GENOSS DES
  <Definition of a complex high-risk patients>
  1. Clinical factors
     * Age 75 or older
     * History of diabetes (those who have had diabetes in the past or are taking diabetes medication)
     * History of chronic kidney disease (GFR <60ml/min/1.73m2) or dialysis
     * History of stroke
     * History of coronary artery bypass graft
     * Left ventricular dysfunction (LVEF <40%)
     * Severe valve disease
     * Acute coronary syndrome with positive troponin levels
  2. Lesion/procedure factors
     * Left main lesion
     * Chronic total occlusion
     * Bifurcation lesion with branches larger than 2 mm
     * Calcified lesion (moderate to severe calcified lesion)
     * Restenosis lesion (in-stent restenosis)
     * Multivessel PCI
     * Three or more stents implanted (≥3 stents implanted)
     * When the stent length of one lesion is more than 50 mm (total stent length >50 mm in a lesion)

SUMMARY:
The objective of study is to evaluate the efficacy and safety of 1 year duration of DAPT after GENOSS® DES Implantation in patients with coronary artery disease according to the complex higher-risk (and indicated) procedure.

DETAILED DESCRIPTION:
The Genoss DES is a novel, biodegradable, polymer-coated, sirolimus eluting stent with a cobalt-chromium stent platform and thin strut. Although the efficacy and safety of this stent have been previously investigated, real-world clinical outcomes data are lacking. Therefore, the objective of this prospective, multicenter study was to evaluate the clinical efficacy and safety of 1 year duration of DAPT after GENOSS® DES Implantation in patients with coronary artery disease according to the complex higher-risk (and indicated) procedure.

The Genoss DES registry is a prospective, single-arm, observational study for evaluation of clinical outcomes of 1 year duration of DAPT after Genoss DES implantation in patients with coronary artery disease according to the complex higher-risk (and indicated) procedure from 9 sites in South Korea. The primary endpoint was a deviceoriented composite endpoint (DOCE), defined as a composite of cardiac death, target vessel-related myocardial infarction (MI), and clinically indicated target lesion revascularization (TLR) at 12 months. The key secondary endpoint was a patient-oriented composite endpoint (POCE), defined as a composite of all-cause death, any myocardial infarction, and any revascularization at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 19 and over
2. Patients with coronary artery disease treated with GENOSS SES
3. Participants who voluntarily decide to participate in this clinical trial, agree to the study protocol and clinical follow-up plan, and provide written informed consent as study participants

Exclusion Criteria:

1. Patients with cardiogenic shock at the time of hospitalization
2. Patients who are pregnant or planning to become pregnant
3. Patients with a life expectancy of less than 1 year
4. Patients participating in randomized controlled trials using other medical devices
5. Patients who have already received treatment with another DES (Drug Eluting Stent) or BMS (Bare Metal Stent) at the time of registration (However, other stent insertions are allowed due to failure of GENOSS DES insertion)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease treated with GENOSS DES
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-oriented composite endpoint | at 12 months after the procedure
  DOCE is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-lesion revascularization (TLR).

SECONDARY OUTCOMES:
Patient-oriented composite endpoint | at 12 months after the procedure
  POCE is defined as a composite of all-cause death, any myocardial infarction, and any revascularization.
All-cause deaths | at 12 months after the procedure
Cardiac death | at 12 months after the procedure
Non-cardiac death | at 12 months after the procedure
Any myocardial infarction | at 12 months after the procedure
Target vessel-realted myocardial infarction (TV-MI) | at 12 months after the procedure
Any revascularization | at 12 months after the procedure
Revascularization of clinically appropriate target lesions | at 12 months after the procedure
Stent thrombosis by ARC definition | at 12 months after the procedure
Lesion success | during the procedure
  When the final residual lesion stenosis is less than 30% using any surgical method.
Procedure success | immediately after the procedure
  When the final residual lesion stenosis is less than 30% using any surgical method, and there is no post-procedure death, myocardial infarction, or revascularization during the hospitalization period.

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon State, South Korea

IPD SHARING:
Plan to Share IPD: No
No The data set is available from the the corresponding author upon reasonable request.